CLINICAL TRIAL: NCT06221306
Title: Radiographic Evaluation of Crestal Bone Loss Around Narrow Diameter Implants Versus Standard Diameter Implants in Conjunction With Bone Augmentation in Horizontally Deficient Posterior Mandibular Partially Edentulous Sites: A Randomized Clinical Trial
Brief Title: Crestal Bone Loss Around Narrow Diameter Implants Versus Standard Diameter Implants With Bone Augmentation in Horizontally Deficient Posterior Mandibular Sites.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Suzy Nabil Naiem, Periodontist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: blt
Record Dates: First submitted 2023-12-17; First posted 2024-01-24 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Horizontal Atrophy of Edentulous Alveolar Ridge

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Narrow diameter implant placement (NDI) (3.3) (Experimental)
  Interventions: Procedure: Dental implant: NDI
- Standard diameter implant (SDI) placement (4.1) with simultaneous bone augmentation. (Active Comparator)
  Interventions: Procedure: Dental implant: SDI

INTERVENTIONS:
Procedure: Dental implant: NDI — Placement of narrow diameter implants (NDI) (3.3) in the dentoalveolar ridge
  Arms: Narrow diameter implant placement (NDI) (3.3)
Procedure: Dental implant: SDI — Placement of standard diameter implants (SDI) (4.1) in the dentoalveolar ridge with simaltenous bone augmentation
  Arms: Standard diameter implant (SDI) placement (4.1) with simultaneous bone augmentation.

SUMMARY:
Dental implant treatment, in many cases, may be impeded by anatomical limitations, such as narrow atrophic ridges. In order to overcome that, additional surgical procedures, such as guided bone regeneration, are often required to augment the deficient hard tissue. However, additional surgical procedures often add morbidity to the patient in addition to prolonging the treatment time and raising the treatment cost.

Hence, simpler, less invasive treatment options are preferred by patients. The use of narrow diameter implants (NDI) offers the great advantage of eliminating the need for augmentation procedures.

DETAILED DESCRIPTION:
Various methods of additional surgical procedures have been introduced to overcome reduced bone volume situations, relevant to the site, size and nature of the defect such as: maxillary sinus floor lifting and augmentation, vertical and lateral ridge augmentation by means of autogenous or bone substitutes, particulate or blocks. Lateral bone augmentation performed simultaneously with implant placement has been a well-established treatment option for horizontal ridge deficiencies.

Such additional procedures are associated with longer surgical time, greater morbidity and greater risk to complications such as: pain, infection, nerve damage, bleeding, wound dehiscence or even graft or implant failure. In addition to, higher treatment cost and a longer healing time. Furthermore, an additional surgical procedure should be considered with caution in medically compromised patients. Moreover, surgical expertise of the operator is required for performing such procedures.

NDIs showed promising results with reported survival rates 95% - 100%. However, prosthetic complications such as: abutment fracture, loss of crown retention and screw loosening were reported.

The successful outcomes of NDI have supported widening the scope to include premolars and molars, particularly where averting an additional augmentation procedure is favoured.

However, areas of concern remain evident regarding; the impact of loading on a reduced surface for osseointegration, the increased probability of fracture, the probable prosthetic complications and the loading stresses affecting crestal bone resorption. In addition to oral health-related quality of life for the patients. Limited literature is found regarding the use of NDI to restore posterior mandibular edentulous sites.

Several studies have compared NDI to SDI in pristine bone. To our knowledge few RCTs compared NDIs to SDI with simultaneous lateral bone augmentation for the treatment of atrophic posterior mandibular ridges, none assessing both crestal bone resorption in addition to oral health related quality of life (OHRQoL) assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients having mandibular edentulous posterior site requiring implant placement.
* Available vertical bone height of ≥ 8 mm in the mandible and ridge width 5-6 mm in width.
* Tooth extraction ≥3 months before surgical intervention.
* Patients without systemic diseases interfering with implant therapy.
* Patients aged ≥ 18 years old.
* Good oral hygiene.

Exclusion Criteria:

* Patients with systemic conditions known to affect bone metabolism and healing
* Patients with habits that may jeopardize the implant longevity and affect the results of the study such as parafunctional habits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Amount of crestal bone changes | 1 year
  Linear measurements (in mm) for the crestal bone level changes on periapical digital radiographs

SECONDARY OUTCOMES:
Prosthetic complications | 1 year
  screw loosening, fracture of restoration

CONTACTS AND LOCATIONS:
Overall Officials: Manal Hosny, Professor, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Greater Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes